CLINICAL TRIAL: NCT05756140
Title: Efficiency of Facial Expression Diagnostic System in Pain Assessment After Geriatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Tülin KURT ALKAN, Doctoral Candidate in Surgical Nursing Science, Zonguldak Bulent Ecevit University
Other Study IDs: 2022-16-09
Record Dates: First submitted 2023-02-16; First posted 2023-03-06 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pain; Aging Problems
Keywords: Geriatric surgery; Pain assessment; Facial diagnosis system
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Group: Geriatric patients in the postoperative period hospitalized in surgical wards
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Control

SUMMARY:
By integrating the methods used in the assessment of pain in geriatric surgery patients with literature, theory and research, this study aims to: evaluate the effectiveness of the facial diagnosis system in the evaluation of pain after geriatric surgery.

The research hypotheses are as follows:

H1: In the evaluation of pain after geriatric surgery, there is a concordance between the pain score evaluated by the patient and the pain score obtained from facial expression diagnostic system analysis.

H1: In the evaluation of pain after geriatric surgery, there is a correlation between the pain score evaluated by the nurse and the pain score obtained from the analysis of the facial expression diagnosis system.

H1: In the evaluation of pain after geriatric surgery, there is a correlation between the pain score evaluated by the patient and the pain score evaluated by the nurse.

DETAILED DESCRIPTION:
By integrating the methods used in the assessment of pain in geriatric surgery patients with literature, theory and research, this study aims to: evaluate the effectiveness of the facial diagnosis system in the evaluation of pain after geriatric surgery.

The number of patients in the groups will be analyzed based on one of the studies to be used in the study. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size is accepted as 0.8, it was seen that at least 68 patients would be sufficient for 80% power. In this way, the criteria sampling method will be used. Anticipated duration is one year.

The inclusion criteria of the patients in the study are as follows:

* The patient is 65 years or older,
* According to the American Society of Anesthesiologists (ASA) classification; Being in class II and III; ASA II: Patient with mild systemic disease, ASA III: Patient with severe systemic disease but not affecting activities of daily living.
* Willingness to participate in the research,
* The patient is awake and oriented after the surgery,
* The patient is not discharged within the first 24 hours after the operation,

Data collecting:

1. An informed consent form will be obtained from patients over 65 years of age in the postoperative period who agreed to participate in the study.
2. Then, the Sociodemographic Data Collection Form created by the researcher will be filled. Sociodemographic form; patient's age, gender, presence of chronic disease, history of surgery, clinical diagnosis of the patient, the patient's surgery, anesthesia during the operation, the patient's ASA score, the nurse's age, the nurse's gender, the nurse's education level, the nurse's clinical experience, the severity of pain felt by the elderly adult patient.
3. After the surgery, when the patient comes to the service and 1 hour after coming to the service, the 3rd and later stages will be repeated. In other words, the patient's pain will be evaluated 2 times in total. The patient and nurse will then be asked to give patient a pain score. Two scales will be used in pain assessment. These are Wong Baker Faces Pain Scale and Numerical Rating Scale.Wong Baker Faces Pain Scale: It consists of 6 different facial expressions, starting with a smiling face and ending with a crying face. Numerical Rating Scale: Patients are asked to draw a number from 0 to 10, 0 to 20, or 0 to 100 that best fits pain intensity. Zero usually indicates "no pain", while the upper limit represents "unbearable pain".
4. And the patient's 30-second facial expression will be recorded with a video camera.
5. This video recording and the score given by the patient will be uploaded to the computer and the pain score.
6. The resulting value will be compared with the value given by the nurses.

ELIGIBILITY:
Inclusion Criteria:

* The patient is 65 years or older,
* According to the American Society of Anesthesiologists (ASA) classification; Being in class -II and III; ASA II: Patient with mild systemic disease, ASA III: Patient with severe systemic disease but not affecting activities of daily living.
* Willingness to participate in the research,
* The patient is awake and oriented after the surgery,
* The patient is not discharged within the first 24 hours after the operation,

Exclusion Criteria:

* Not being willing to participate in the research,
* The presence of any facial anomalies that may change the facial expression analysis of the patient,
* The patient's regular use of opiates in the last 6 months,
* The patient has undergone surgical intervention that requires not being in the prone or semifowler position,
* The patient is not awake and oriented after the surgery,
* Discharge of the patient within the first 24 hours after surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The research sample will consist of geriatric patients aged 65 and over who were hospitalized in the post-operative general surgery service.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Determination of the average scores from the "Wong Baker Facial Pain Scale" | 6 months
  Wong Baker Facial Pain Scale: It consists of 6 different facial expressions, starting with a smiling face and ending with a crying face. The patient and the nurse will be asked to give a pain score to the patient when immediately after the patient comes from the surgery and 1 hour after coming to the service.
Determination of the average scores from the "Numerical Rating Scale" | 6 months
  Numerical Rating Scale: Patients are asked to draw a number from 0 to 10, 0 to 20, or 0 to 100 that best fits pain intensity. Zero usually indicates "no pain", while the upper limit represents "unbearable pain". The patient and the nurse will be asked to give a pain score to the patient when immediately after the patient comes from the surgery and 1 hour after coming to the service.

SECONDARY OUTCOMES:
Machine learning will be provided using a computer-assisted facial expression recognition system. | 12 months
  The 30-second facial expression of the patient is recorded with a video camera immediately after the patient leaves the surgery and comes to the service and 1 hour after coming to the service. With this video recording and the score given by the patient, the pain score will be uploaded to the computer. The obtained value will be compared with the value given by the nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Tülin KURT ALKAN, Expert, Principal Investigator — https://zonguldakataturkdh.saglik.gov.tr/?_Dil=1
Locations (1):
- Zonguldak Ataturk State Hospital, Zonguldak, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kur Alkant T, Tasdemir N. Testing Machine Learning-Based Pain Assessment for Postoperative Geriatric Patients. Comput Inform Nurs. 2025 Nov 1;43(11):e01248. doi: 10.1097/CIN.0000000000001248. PMID 39761361